CLINICAL TRIAL: NCT06557993
Title: Effectiveness of Serratus Posterior Superior Intercostal Plane Block Applied With Ultrasonography in Myofascial Pain Syndrome
Status: Recruiting | Type: Observational
Sponsor: Halil Ibrahim Altun (Other)
Responsible Party: Sponsor-Investigator, Halil Ibrahim Altun, pain specialist, Kanuni Sultan Suleyman Training and Research Hospital
Organization: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Other Study IDs: MyofascialPainSyndrome
Record Dates: First submitted 2024-08-12; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Pain, Neck
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Serratus Posterior Superior Intercostal Plane Block — The serratus posterior superior muscle is located deep to the rhomboid major and minor. Ligamentum nuchae starts from the processus spinosus of C7-T3 vertebrae and extends to the 2nd-5th. In the ribs, the angulus ends at the upper edge of the rib. Serratus posterior superior -intercostal plane block (SPSİPB) is a newly defined block, and C7-T7 spread has been shown in cadaver studies

SUMMARY:
Trigger point treatment in myofascial pain syndrome should be planned according to its etiology to prevent relapses. Although there are various modalities, in cases where medical and noninvasive methods are ineffective, diluted local anesthetic injections or diluted local anesthetic injections with steroids, and sometimes dry needling or botulinum toxin, are preferred. In recent years, imaging methods such as ultrasonography have been frequently used for trigger point injections. These injections may be repeated for several sessions depending on the patient's response. Pain, local anesthetic toxicity, bleeding, allergic reactions, pneumothorax, intramuscular hematoma, cerebrovascular events, spinal injury, vasovagal syncope and infections have been reported during injections. Therefore, during trigger point injections, vascular access should be established in the patient, the patient should be monitored, injections should be performed under sterile conditions, and an emergency kit should be kept ready in all cases .

The serratus posterior superior muscle is located deep to the rhomboid major and minor. Ligamentum nuchae starts from the processus spinosus of C7-T3 vertebrae and extends to the 2nd-5th. In the ribs, the angulus ends at the upper edge of the rib. Serratus posterior superior -intercostal plane block (SPSİPB) is a newly defined block, and C7-T7 spread has been shown in cadaver studies . In our study, investigators compared the newly defined SPSİPB, which is practical to be applied with USG in Myofascial Pain Syndrome (MAS), which is frequently seen especially in young people and desk workers, with trigger point injection, which has been used in the treatment of MAS for many years and whose effectiveness has been proven, and SPSİPB applied from a single point with USG guidance. investigators aimed to contribute to the literature regarding the effectiveness of in MAS. The newly defined rhomboid intercostal plane block and SPSIPB are routinely applied successfully in our algology clinic in patients with MAS and postzoster neuralgia in the thoracic region.

DETAILED DESCRIPTION:
Myofascial Pain Syndrome is a condition characterized by sensory, motor and autonomic symptoms caused by trigger points (TN), which have a source of pain within the muscle and fascia. Trigger points are hyperirritable points located within taut bands. The aim of the treatment is to inactivate trigger points and relax tense muscle bands. The goal is to eliminate muscle tension and achieve normal muscle length, function and strength. Needling methods are still considered the most effective method in the initial treatment of MAS. Local anesthetic (LA) injection is a frequently used method with proven effectiveness .

Although the etiology of the ethical points accompanying MAS has not been elucidated; It is thought that posture disorders, vitamin-mineral deficiencies, metabolic diseases, genetic factors, stress and overuse disrupt the contraction-relaxation cycle in muscle sarcomeres. An acidic and hypoxic environment occurs in the muscle, inflammatory mediators are released, and this situation is more common in phasic muscles than in tonic muscles. Trigger points are divided into two: active and latent. In active trigger points, the patient's complaint is triggered by palpation and a jump sign is obtained, while in latent trigger points, pain occurs with palpation, but the patient's complaint is not triggered. During the examination, the trigger point is compressed and a local twitch response is obtained. Sometimes trigger points can also cause autonomic symptoms and referred pain .

The study was conducted at the Algology Department of Kanuni Sultan Süleyman Training and Research Hospital, between March 2023 and March 2024, on patients aged 18-65 who had MAS and therefore had serratus posterior superior intercostal plane block or trigger point injection applied to the neck-back region in a single session. It will be done by retrospectively scanning the files of the patients . Within the scope of the research, age, gender, Visual Analog Scale (VAS), Neck disability scores and Algometric measurements before and in the first and third months after the procedure will be scanned from patient files and those that can be accessed will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65 and having been diagnosed with MAS based on the MAS diagnostic criteria,
* No invasive procedure has been performed for this disease in the last 3 months
* Signing the informed consent form
* Patients with complete data to be scanned in their files

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Cervical disc herniation,
  * history of trauma/operation to the neck,
  * shoulder or back area, malignancy, presence of kyphoscoliosis,
  * inflammatory diseases (rheumatoid arthritis, ankylosing spondylitis, etc.),
  * congenital anomalies of the spine, neck pain accompanied by neurological deficit,
  * pregnancy, mental or psychotic disorder, bleeding and Hematological diseases that cause coagulation disorders, use of antiplatelet, anticoagulant and drugs that cause bleeding tendencies, serious systemic and local infection in the intervention area such as sepsis, and allergy to any of the drugs to be used.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
onset of pain and application time of intervention Visual Analog Scale (VAS) | four months

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No